CLINICAL TRIAL: NCT03972956
Title: Samples Procurement for Patients With Colorectal Cancer, Gastric Cancer, and Non-malignant Disease Undergoing Surgery
Brief Title: Samples Procurement for Colorectal Cancer, Gastric Cancer, and Non-malignant Disease
Status: Recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Tao Fu, Director of Department of GI Surgery II, Renmin Hospital of Wuhan University
Other Study IDs: SAMPGICUS
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer; Gastric Cancer; Inflammatory Bowel Diseases; Gastric Ulcer; Hemorrhoids; Hernia
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Inflammatory Bowel Diseases; Stomach Ulcer; Hemorrhoids; Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens will be analyzed to study, but not limited to, genomics, epigenomics, and proteomics.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal cancer or gastric cancer patient: Patients suffering from CRC or gastric cancer scheduled to have surgical resection of colon/rectum or stomach.
  Interventions: Other: No intervention will be given to patients.
- Non-malignant disease patient: Patients suffering from non-malignant disease scheduled to have surgery.
  Interventions: Other: No intervention will be given to patients.

INTERVENTIONS:
Other: No intervention will be given to patients. — Samples are collected at the time of a scheduled surgery that is part of normal treatment. This study will not have any impact on the care or treatment the patient receives.

SUMMARY:
The purposes of this study are to collect and store samples including blood, normal and tumor tissue from patients with colorectal cancer or gastric cancer, to collect and store samples including blood and/or normal gastrointestinal tissue (if available) from patients with non-malignant disease (including, but not limited to, inflammatory bowel disease (IBD), gastric ulcer, hemorrhoids or hernia), and to create a database for the collected samples and allow access to relevant clinical information for current and future protocols.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with colorectal cancer, gastric cancer, non-malignant disease that requires undergoing surgery.
* Must be willing and able to provide informed consent.

Exclusion Criteria:

* Subjects whose comorbidities would preclude diagnostic or therapeutic intervention.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who are planning to undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Confirmation of diagnosis by pathologist | Up to 3 years
  Once tissue is collected, those samples that have a confirmed diagnosis of disease by the pathologist will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Fu, MD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Department of Gastrointestinal Surgery II, Renmin Hospital of Wuhan University, Wuhan, Hubei, China